CLINICAL TRIAL: NCT01563068
Title: A Phase 1, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of Calcipotriene Foam, 0.005%, Applied Under Maximal-Use Conditions in Adolescent Subjects (Ages 12 to 16 Years) With Plaque Psoriasis
Brief Title: Safety, Tolerability, PD & PK of Calcipotriene 0.005% Foam, Under Maximal Use in 12-16 Year Olds With Plaque Psoriasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayne Pharma International Pty Ltd (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STF115750
Record Dates: First submitted 2012-03-15; First posted 2012-03-26 (Estimated); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Psoriasis
Keywords: plaque psoriasis; pediatric; adolescent
MeSH Terms: conditions — Psoriasis | interventions — calcipotriene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (1):
- Calcipotriene Foam (Experimental): Calcipotriene foam 0.005% administered under maximal-use conditions to adolescent patients with plaque psoriasis
  Interventions: Drug: Calcipotriene 0.005% Foam

INTERVENTIONS:
Drug: Calcipotriene 0.005% Foam — Topical application applied twice a day for 15 days
  Other Names: Sorilux

SUMMARY:
Calcipotriene is a vitamin D3 analog that has been used as topical therapy in adult subjects with plaque-type psoriasis since 1993. Calcipotriene foam, 0.005%, was approved in 2010 for the treatment of plaque psoriasis in adults aged 18 years and older. The current study is a multicenter study in which adolescent subjects (ages 12 to 16 years, inclusive) or their primary caregivers will apply calcipotriene foam, 0.005%, as a thin layer to treatment areas of the body and scalp, excluding the face, under maximal use conditions, twice a day for 14 days and once on Day 15. The safety, tolerability, pharmacodynamics, and pharmacokinetics of calcipotriene will be evaluated

DETAILED DESCRIPTION:
This Phase 1 multicenter, open-label, repeat-dose study is designed to evaluate the safety, tolerability, pharmacodynamics, and pharmacokinetics of calcipotriene foam, 0.005%, applied topically to adolescent subjects with moderate plaque psoriasis (defined as a score of 3 on the Investigator's Static Global Assessment [ISGA]) involving a minimum of 10% body surface area (BSA) excluding the face and scalp, and a minimum of 20% scalp involvement. Subjects will be enrolled no more than 2 weeks after Screening. Approximately 30 eligible subjects, ages 12 to 16 years, inclusive, will be enrolled to ensure 20 completing subjects. Calcipotriene foam will be applied as a thin layer twice a day for 14 days and once on Day 15 on all treatment areas. Blood samples for the evaluation of albumin adjusted calcium, intact parathyroid hormone (iPTH), alkaline phosphatase, magnesium, and phosphorus will be taken at Screening and on Day 1 (before the first dose), Day 15 (3 to 9 hours after dosing), and on Day 22 if the results from Day 15 show any abnormalities. Serum 25-OH vitamin D concentrations will be evaluated on Day 1 (before the first dose). Safety and tolerability will be evaluated throughout the treatment period and a 7 day follow-up period. Blood samples for pharmacokinetic (PK) evaluation will be collected on Days 1 and 15. Urine samples for evaluation of calcium/creatinine ratio will be collected before dosing on Days 1 and 15.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, ages 12 to 16 years, inclusive, at the time of consent.
2. Plaque psoriasis involving 10% body surface area (excluding the scalp and face).
3. 20% scalp involvement (excluding the body and face).
4. Clinical diagnosis of mild to moderate plaque psoriasis, as defined by an ISGA score at Screening of 3 on a scale of 0 to 4.
5. The ability and willingness of the subject and the subject's primary caregiver to follow all study procedures, attend all scheduled visits, and successfully complete the study.

5. The subject's parent(s) or legal guardian must have the ability to understand and sign a written informed consent form and a Health Insurance Portability and Accountability Act (HIPAA) authorization form, which must be obtained prior to participation in this study. The HIPAA authorization may be incorporated in the informed consent form. Also, the subject's assent must be obtained and documented.

Exclusion Criteria:

1. Any inflammatory skin disease in the treatment area that may confound the evaluation of the plaque psoriasis (eg, atopic dermatitis, contact dermatitis, tinea corporis).
2. Current diagnosis of unstable forms of psoriasis in the treatment area, including guttate, erythrodermic, exfoliative, or pustular psoriasis.
3. Use of any topical product (including sunscreen, creams, ointments, lotions, and powders) applied on or near the treatment area within 48 hours prior to enrollment.
4. Use of topical treatments that have a known beneficial effect on psoriasis, including but not limited to corticosteroids, retinoids, vitamin D derivatives, coal tar, tazarotene, or anthralin, medicated shampoos within 2 weeks prior to enrollment.
5. Use of nonbiologic systemic antipsoriatic therapy (eg, corticosteroids, retinoids, methotrexate, cyclosporine, other immunosuppressive agents), biologic therapy (eg, alefacept, etanercept, efalizumab), or phototherapy (eg, ultraviolet A, psoralen and ultraviolet A, ultraviolet B) within 4 weeks prior to enrollment.
6. Use or need for initiation of any nonpsoriatic therapy that might affect psoriasis (including antimalarials, adrenergic receptor blockers, interferon, or lithium) within 4 weeks prior to enrollment.
7. Use of medications that affect or change calcium and parathyroid hormone (PTH) concentrations or interfere with the measurement of calcium or PTH concentrations within 4 weeks prior to enrollment.
8. Known difficult venous access beyond that expected for subject age.
9. Any serious skin disorder or any chronic medical condition that is not well controlled.
10. Positive urine drug screen result for alcohol, cotinine, or drugs of abuse at the time of Screening.
11. Average daily ingestion of more than 2000 mg of elemental calcium or more than 1000 IU of vitamin D within 2 weeks prior to enrollment.
12. Current drug or alcohol abuse.
13. History of hypersensitivity, known allergy, or other adverse reaction to calcipotriene or other vitamin D analogs or to any component of the study product.
14. Current or past history of hypercalcemia, vitamin D toxicity, severe renal insufficiency, or severe hepatic disorders.
15. Use of any investigational therapy within 4 weeks prior to enrollment.
16. Pregnant, breastfeeding, or sexually active female subjects of childbearing potential (after menarche) who are not practicing an acceptable method of contraception. Acceptable methods of contraception include one of the following highly effective methods of contraception (ie, Pearl Index <1.0%): complete abstinence from intercourse or 2 forms of barrier contraception (diaphragm plus spermicide for females, condom plus spermicide for males), or systemic contraceptives (combined or progesterone only) used in combination with a condom. The subject must agree to use an acceptable method of contraception from 2 weeks prior to administration of study product, throughout the study, and for 28 days after completion or premature discontinuation from the study.
17. Current immunosuppression.
18. Albumin-adjusted serum calcium at Screening that is outside the normal reference range.
19. Any other condition that, in the judgment of the investigator, would put the subject at unacceptable risk for participation in the study.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Effect of calcium metabolism | Up to 3 Weeks
  determine albumin-adjusted calcium, iPTH, alkaline phosphatase, and phosphorus

SECONDARY OUTCOMES:
Pharmacokinetics | predose, 1,2,3,4,6 hours postdose
  Area Under Curve (AUC)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Investigational Site, San Diego, California
  - Investigational Site, Ormond Beach, Florida
  - Investigational Site, Tampa, Florida
  - Investigational Site, Marietta, Georgia
  - Investigational Site, Chicago, Illinois
  - Investigational Site, Indianapolis, Indiana
  - Investigational Site, Louisville, Kentucky
  - Investigational Site, Philadelphia, Pennsylvania
  - Investigational Site, Houston, Texas